CLINICAL TRIAL: NCT02870803
Title: OCT-angiography in Diabetic Patients: Qualitative Changes of the Intermediate and Deep Capillary Plexuses After Resolution of Macular Edema by Intravitreal Pharmacotherapy
Brief Title: OCT-angiography in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Retina Clinic, Sao Paulo, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: Retina Clinic / OCT
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Around the world there is an increasing incidence of diabetes mellitus, with millions of people affected. In this population, diabetic macular edema (DME) is the most common cause of visual impairment. While the visual impairment caused by EMD is variable, its early treatment can improve visual acuity and quality of life. The objective of this project is to use the new OCT-angiography technology, which evaluates macular capillary network without the need of intravenous injection of contrast, to assess macular microcirculatory network in its response to intravitreal pharmacological treatment of EMD. The resulting qualitative evaluation can be helpful in understanding the pathophysiology of visual loss associated with DME and in determining prognosis.

DETAILED DESCRIPTION:
Patients who participate in this study will be selected among adults treated at the Retina Clinic and Ocular Oftalmologia clinics and will be aware of all stages of the research, formalizing the approval of their participation by informed consent term. The tests will be performed after pupillary dilation with 2 eye drops of tropicamide 1% (Mydriacyl, Alcon Laboratories), in Cirrus 5000 HD-OCT devices (Carl Zeiss Meditec - Dublin USA). Image acquisition protocols Optic Disc Cube 200x200 and 512x128 Macular Cube will be used, with analysis by RNFL protocols and NGO Analysis Report and Macular Cube Analysis Report, respectively. Subjective analysis of the examinations will be performed by the three authors of this project independently and then compared between them.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of diabetes mellitus type 1 or 2;
* Age equal or greater than 18 years;
* At least one eye with diabetic macular edema and central thickness greater than or equal to 290 microns (female patients) or 305 microns (males) measured by OCT and subjected to intravitreal pharmacotherapy.

Exclusion Criteria:

* Aphakic patients;
* History of major eye surgeries (vitrectomy, cataract surgery, scleral buckle, other intraocular surgery) in the last 4 months;
* Tractional retinal detachment involving the macula, vitreomacular traction syndrome or other concurrent macular diseases;
* Advanced or uncontrolled glaucoma (according to the investigator's judgment); Evidence of angle neovascularization;
* Presence of an eye condition (besides diabetic retinopathy) which, in the opinion of the investigator, may alter the visual acuity during the study course (e.g. venous or arterial retinal occlusions, uveitis or other ocular inflammatory diseases, neovascular glaucoma, etc.);
* Significative cataract which, in the opinion of the investigator, may be decreasing visual acuity in 3 lines or more;
* History of YAG Laser capsulotomy in the last 2 months;
* Severe renal disease, defined as chronic renal failure requiring dialysis or a kidney transplant;
* Blood pressure higher than 180/110 mmHg, acute myocardial infarction, other acute cardiac events requiring hospitalisation, stroke, transient ischemic attack or treatment for congestive heart failure;
* Systemic treatment with anti-VEGF or pro-VEGF in the last 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic macular edema.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-11 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
OCT-angiography qualitative changes | 12 months
  Assess the OCT-angiography qualitative changes observed in intermediate and deep capillary networks in diabetic patients after the resolution of macular edema with intravitreal drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: André Maia, M.D., Study Chair — Retina Clinic CEO
Locations (1):
- Retina Clinic, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klein R, Klein BE, Moss SE. Visual impairment in diabetes. Ophthalmology. 1984 Jan;91(1):1-9. PMID 6709312
- [Result] Kiri A, Dyer DS, Bressler NM, Bressler SB, Schachat AP. Detection of diabetic macular edema: Nidek 3Dx stereophotography compared with fundus biomicroscopy. Am J Ophthalmol. 1996 Nov;122(5):654-62. doi: 10.1016/s0002-9394(14)70483-0. PMID 8909204
- [Result] Puliafito CA, Hee MR, Lin CP, Reichel E, Schuman JS, Duker JS, Izatt JA, Swanson EA, Fujimoto JG. Imaging of macular diseases with optical coherence tomography. Ophthalmology. 1995 Feb;102(2):217-29. doi: 10.1016/s0161-6420(95)31032-9. PMID 7862410
- [Result] Knudsen ST, Bek T, Poulsen PL, Hove MN, Rehling M, Mogensen CE. Macular edema reflects generalized vascular hyperpermeability in type 2 diabetic patients with retinopathy. Diabetes Care. 2002 Dec;25(12):2328-34. doi: 10.2337/diacare.25.12.2328. PMID 12453981
- [Result] Ozdek SC, Erdinc MA, Gurelik G, Aydin B, Bahceci U, Hasanreisoglu B. Optical coherence tomographic assessment of diabetic macular edema: comparison with fluorescein angiographic and clinical findings. Ophthalmologica. 2005 Mar-Apr;219(2):86-92. doi: 10.1159/000083266. PMID 15802932
- [Result] Otani T, Kishi S. Correlation between optical coherence tomography and fluorescein angiography findings in diabetic macular edema. Ophthalmology. 2007 Jan;114(1):104-7. doi: 10.1016/j.ophtha.2006.06.044. Epub 2006 Oct 27. PMID 17070586